CLINICAL TRIAL: NCT00026754
Title: Eligibility Screening for the NIH Intramural Research Program Clinical Protocols
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010129; 01-C-0129
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Sarcoma; Melanoma
Keywords: Screening; Cancer; HIV Infection; Scans; Laboratory Tests; HIV; Skin Disorders
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Sarcoma; Melanoma; Neoplasms; HIV Infections; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients
- Cohort 2: Healthy Volunteers

SUMMARY:
The purpose of this protocol is to provide patients with adequate informed consent to understand that screening tests with minimal health risk will be performed to evaluate their eligibility for a research study. The protocol makes it clear that patients initial visit to the intramural clinical program may include screening studies that are not medically necessary for disease management, but are done purely for research purposes.

Patients with a known or suspected diagnosis of cancer, HIV infection, skin disorder or immunodeficiency who are being considered for enrollment in a National Cancer Institute intramural clinical research protocol will participate in this consent protocol. It informs patients of screening tests and procedures involving minimal risk that are done for research purposes only, including blood tests, electrocardiogram, standard X-rays (e.g., chest X-ray), bone films, computed tomography (CT), magnetic resonance imaging (MRI), and nuclear medicine studies. It explains that other eligibility screens that are more invasive and involve greater risk, such as a biopsy, will require separate consent.

...

DETAILED DESCRIPTION:
Background:

Patients and healthy volunteers who are being evaluated for NIH Intramural Research Program (IRP) protocols must be screened to determine whether they meet the eligibility criteria prior to enrollment.

Objectives:

Evaluate patient or healthy volunteer eligibility for participation in NIH IRP research protocols.

Collect results of screening test for use on subsequent research protocols as baseline (e.g., pretreatment) values.

Collect specific research samples required for the primary research protocol as part of a screening test or procedure in order to avoid from having to subject the patient to a painful procedure on multiple occasions.

Eligibility:

Patients and healthy volunteers who are being evaluated for and treated on protocols within the NIH IRP.

Design:

This protocol is not a research study of an investigational drug or device.

Screening tests and procedures that are required by the primary research protocols are conducted in order to establish eligibility for these protocols.

In some cases, specific research samples required for the primary research protocol may be collected during the screening process in order to avoid from having to subject the patient to a painful procedure on multiple occasions.

Tissues and biological fluids that are obtained during the screening process will be stored.

Once a patient or healthy volunteer completes the screening process and is either enrolled onto another NIH study or is returned to the care of their local physician they will be taken off study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients and healthy volunteers who are being evaluated for protocols within the NIH Intramural Research Program (IRP). Note: Participants must be > 1 month of age.
* All patients or their parent/guardians or Legally Authorized Representative (LAR) must sign a document of informed consent indicating their understanding of the research nature and the risks of the procedures that will be performed to assess eligibility for research protocols. NOTE: It is expected that healthy adult volunteers have the capacity to consent (i.e., a LAR may not be used).

EXCLUSION CRITERIA:

None

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and healthy volunteers who are being evaluated for NIH Intramural Research Program (IRP) protocols must be screened to determine whether they meet the eligibility criteria prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 19522 (Actual)
Dates: Start 2004-01-14 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Tissue for future research | 10 years
  Tissue remaining from collections during the screening process, either for research eligibility or as clinically indicated may be stored for future research
Screening testing/results | 10 years
  Collect results of screening test for use on subsequent research protocols as baseline (e.g., pretreatment) values
Research sample collection | 10 years
  Collect specific research samples required for the primary research protocol as part of a screening test or procedure in order to avoid from having to subject the patient to a painful procedure on multiple occasions
Numbers of screened patients and healthy volunteers | 10 years
  Gather prospective information on the number of patients screened for a particular study and compare to those enrolled onto an interventional study or natural history study.
Eligibility evaluations | 10 years
  Evaluate patient eligibility for participation in NCI/CCR research protocols

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0129.html